CLINICAL TRIAL: NCT02476448
Title: Evaluation of Ureteral Jets on Cystoscopy: A Randomized Controlled Trial
Brief Title: Evaluation of Ureteral Jets on Cystoscopy
Acronym: JET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cecilia Calvo (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Cecilia Calvo, Quality Assurance, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FLA 15-015
Record Dates: First submitted 2015-02-24; First posted 2015-06-19 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Injury of Ureter
Keywords: ureteral jet; pelvic surgery; cystoscopy
MeSH Terms: interventions — Saline Solution; Sodium Chloride; Phenazopyridine; Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal Saline (Active Comparator): Infused into the bladder to allow for visualization of bladder walls and urine jets.
  Interventions: Drug: Normal saline
- Dextrose 10% (Experimental): Infused into the bladder to allow for visualization of bladder walls and colored urine jets.
  Interventions: Drug: Dextrose 10%
- Phenazopyridine (Experimental): Will be administered (orally) preoperatively and will be evaluated for its colorization properties during cystoscopy.
  Interventions: Drug: Phenazopyridine
- Sodium Fluorescein (Experimental): Will be administered (intravenously) prior to the cystoscopy and will be evaluated for its colorization properties during cystoscopy.
  Interventions: Drug: Sodium Fluorescein

INTERVENTIONS:
Drug: Normal saline — Used to distend the bladder for cystoscopic evaluation
  Other Names: Saline; NS
  Arms: Normal Saline
Drug: Phenazopyridine — Administered orally preoperatively and assessed during cystoscopy
  Other Names: Pyridium; AZO
  Arms: Phenazopyridine
Drug: Dextrose 10% — Used to distend the bladder for cystoscopic evaluation
  Other Names: D10
  Arms: Dextrose 10%
Drug: Sodium Fluorescein — Administered intravenously and assessed during cystoscopy
  Other Names: Fluorescein; Fluorocyte
  Arms: Sodium Fluorescein

SUMMARY:
This study evaluates 4 different methods to aid surgeons to visualize ureteral jets on cystoscopy.

DETAILED DESCRIPTION:
This study proposes to test and compare the surgeon's impression/confidence in identifying ureteral jets using 3 other methods in contrast to standard diagnostic cystoscopy: 1) cystoscopy with Dextrose 10% solution, 2) cystoscopy with phenazopyridine and 3) IV sodium fluorescein 4) standard cystoscopy with saline.

ELIGIBILITY:
Inclusion Criteria:

* adult
* undergoing a cystoscopy or as part of their planned procedure

Exclusion Criteria:

* Chronic kidney disease
* known prior surgical removal of kidney or ureteral obstruction
* Current ureteral stent placed
* Allergy to any of the interventions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Davila, MD, Study Chair — Cleveland Clinic Florida; Alexandriah Alas, MD, Study Director — Cleveland Clinic Florida; Luis M Espaillat, MD, Principal Investigator — Cleveland Clinic Florida; Eric A Hurtado, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espaillat-Rijo L, Siff L, Alas AN, Chadi SA, Zimberg S, Vaish S, Davila GW, Barber M, Hurtado EA. Intraoperative Cystoscopic Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1378-1383. doi: 10.1097/AOG.0000000000001750. PMID 27824741

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenazopyridine: Will be administered (PO) preoperatively and will be evaluated for its colorization properties during cystoscopy.
  Phenazopyridine: Administered orally preoperatively and assessed during cystoscopy
- Sodium Fluorescein: Will be administered (IV) prior to the cystoscopy and will be evaluated for its colorization properties during cystoscopy.
  Sodium Fluorescein: Administered intravenously and assessed during cystoscopy
Period: Overall Study
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein
Started | 44 (one given phenazopyridine pre-op and was analyzed in her randomization group per intention to treat) | 44 | 44 | 44
Completed | 44 | 44 | 44 | 44
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein | Total
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (13.8) | 59.3 (12.1) | 60 (9.7) | 60.3 (13.9) | 60.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 44 | 44 | 176
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Full Range); unit: kg/m^2] | 26.4 [19.8 to 38.9] | 26.9 [22.1 to 38.8] | 30.3 [21.6 to 41.0] | 26.7 [20.6 to 42] | 27.6 [19.8 to 42]

OUTCOME MEASURES:

1. Primary Outcome: Ureteral Jet Visibility
Description: Surgeons will chose from a likert scales as either:
  1. not visible
  2. Somewhat visible
  3. clearly visible This will be completed during the cystoscopic evaluation
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein
Number analyzed (Participants) | 44 | 44 | 44 | 44
Participants
  Clearly Visible | 22 | 35 | 27 | 41
  Somewhat Visible | 17 | 9 | 16 | 3
  Not Visible | 5 | 0 | 1 | 0

2. Secondary Outcome: Surgeon Satisfaction
Description: A 4 point likert scale will be completed during the procedure to assess satisfaction as follows:
  1. very satisfied
  2. satisfied
  3. somewhat satisfied
  4. unacceptable
Time Frame: 5 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein
Number analyzed (Participants) | 44 | 44 | 44 | 44
Participants
  Very Satisfied | 12 | 27 | 12 | 26
  Satisfied | 14 | 12 | 15 | 13
  Somewhat Satisfied | 13 | 5 | 12 | 4
  Unacceptable | 5 | 0 | 5 | 1

3. Other Pre Specified Outcome: Number of Participants With Urinary Tract Infections
Description: Medical records will be followed prospectively for 6 weeks to assess for incidence of urinary tract infections within different groups.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein
Number analyzed (Participants) | 44 | 44 | 44 | 44
Participants | 10 | 13 | 9 | 10

ADVERSE EVENTS:
Arm/Group | Normal Saline | Dextrose 10% | Phenazopyridine | Sodium Fluorescein
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/44 | 1/44 | 0/44 | 1/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline (N=44) | Dextrose 10% (N=44) | Phenazopyridine (N=44) | Sodium Fluorescein (N=44)
Elevated blood pressure (Cardiac disorders) | 1 | 0 | 0 | 0
parathesia (Nervous system disorders) | 1 | 0 | 0 | 0
chest pain (Cardiac disorders) | 0 | 1 | 0 | 0
Post-op retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 — W/ bladder rupture POD#4

LIMITATIONS AND CAVEATS:
Weaknesses include that without any postoperative diagnoses of ureteral injury, we cannot comment on the sensitivity or specificity of each method.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No